CLINICAL TRIAL: NCT03892525
Title: Phase Ib Study Evaluating the Safety and Efficacy of Intratumoral Agonistic Anti-CD40 (Selicrelumab) in Combination With Anti-PDL1 (Atezolizumab) in Patients With Refractory or Relapsed B Cell Lymphoma
Brief Title: Study of Intratumoral Selicrelumab With Atezolizumab in Patients With Refractory or Relapsed B Cell Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: End of drug development
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ITSELF
Record Dates: First submitted 2019-03-26; First posted 2019-03-27 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Recurrent B-Cell Non-Hodgkin Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — selicrelumab; atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental)
  Interventions: Drug: Selicrelumab; Drug: Atezolizumab

INTERVENTIONS:
Drug: Selicrelumab — escalated dose in intratumoral injection, every 3 weeks, for 3 cycles
Drug: Atezolizumab — 1200mg IV every 3 week until progression or relapse for maximum 1 year
  Other Names: Tecentriq

SUMMARY:
This is a multicenter, open, dose escalation phase Ib trial of intratumoral agonistic anti-CD40 Ab (Selicrelumab intratumoral every 3 weeks for 3 cycles) in combination with anti-PDL1 Ab (Atezolizumab 1200mg intravenous every 3 weeks) in patients with refractory or relapsed B cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 and older
2. Histologically confirmed diagnosis of recurrent or refractory B-non-Hodgkin's lymphoma (NHL)
3. At least one injectable lesion:

   i) at least one nodal lesion amenable to intratumoral injection and biopsy (including deep lesions accessible by interventional radiology either under US or CT-scan guidance). The first injected lesion should be of at least 2 x 1.5 cm in diameter. The subsequent lesions to be injected should be ≥1.5 cm in diameter. Extra nodal lesions will not be considered as injectable lesion.

   ii) OR One cutaneous lesion of at least ≥ 1 cm in diameter. Other extra nodal lesion will not be considered as injectable lesion.
4. Patient must have a 18-F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose (FDG) avid lymphoma that can be followed by positron emission tomography (PET).
5. Bi-dimensionally measurable disease defined by at least one measurable lesion according to Lugano criteria, with at least 1cm in its shortest diameter and 1.5cm in largest diameter (different from the lesion that will be injected)
6. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1
7. Signed written informed consent
8. Life expectancy ≥ 3 months
9. Patients must have recovered to ≤ grade 1 from all toxicities related to prior treatments excluding alopecia.
10. Patients must be naïve from immunotherapy with anti-PD1/PDL1 or agonistic anti-CD40 therapy
11. Adequate laboratory parameters:

    * Hb ≥ 9 g/dl
    * absolute neutrophil count (ANC) ≥ 1000/μL
    * Platelet count ≥ 50,000/μL
    * Total bilirubin < 2.5 times the institutional upper limit of normal (ULN) (3.5 x ULN if liver involvement)
    * Hepatic enzymes (aspartate aminotransferase (AST), alanine aminotransferase (ALT) ) ≤ 2.5 x ULN (5 x ULN if liver involvement)
    * Serum creatinine < 2.0 x ULN or creatinine clearance >50 mL/mn
    * International Normalized Ratio (INR) and Partial Thromboplastin Time (PTT) >1.5 × ULN
12. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 72 hours prior to the start of study drug administration.
13. Persons of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 6 months after study drug is stopped.

    *Highly effective method includes: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation 1 (oral/ intravaginal/ transdermal); progestogen-only hormonal contraception associated with inhibition of ovulation 1 (oral/injectable/implantable); intrauterine device (IUD); intrauterine hormone-releasing system (IUS); bilateral tubal occlusion; vasectomised partner; sexual abstinence
14. Patient covered by any social security system (France)
15. Patient who understands and speaks one of the country official language

Exclusion Criteria:

1. Immature B cell malignancies (B-acute lymphoblastic leukemia (ALL), Burkitt lymphoma) and T-cell lymphomas
2. History of severe allergic anaphylactic reactions to chimeric, human or humanized antibodies, or fusion proteins or known hypersensitivity to Chinese hamster ovarian (CHO) cell products or any component of the Atezolizumab formulation. Patients with a known allergy to either of the drugs individually
3. Use of any standard or experimental anti-cancer drug therapy within 4 weeks prior to the first scheduled treatment dose (C1D1).
4. History of treatment with anti-PD1 or anti-PDL1.
5. Significant immunosuppression from:

   * Concurrent, recent (≤ 2 weeks ago) or anticipated treatment with systemic corticosteroids at dose >10mg/day of prednisolone (or equivalent)
   * Other immunosuppressive medications such as methotrexate, cyclosporine, azathioprine
   * Any immunosuppressive condition such as common variable hypogammaglobulinemia
6. Myocardial infarction within 6 months prior to first study drug, active cardiac ischemia or New York Heart Association (NYHA) Grade III or IV heart failure, severe arrhythmia, unstable arrhythmias, or unstable angina) or pulmonary disease (including uncontrolled obstructive pulmonary disease and history of bronchospasm or other according to investigator's decision)
7. left ventricular ejection fraction (LVEF) < 45% as determined by echocardiography or multiple uptake gated acquisition (MUGA) scan
8. Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
9. Prior history of other cancer other than lymphoma within 2 years (except basal cell carcinoma, in situ squamous and non-squamous cell carcinomas completely resected (R0) and prostate cancers with normal results for more than 6 months)
10. Recent (< 1 month ago) clinically significant infection, active tuberculosis or antibiotics therapy
11. Central nervous system involvement with lymphoma, including parenchymal and leptomeningeal disease. Patients with asymptomatic focal epiduritis on imaging might be included with the Sponsor's approval.
12. Ongoing or history of autoimmune disease, including active non-infectious pneumonitis, with the exception of alopecia, vitiligo, auto-immune endocrine deficiency with stable hormone replacement therapy, controlled skin eczema and stable asymptomatic and treated asthma. Patients with severe auto-immune disease in one of their parents, siblings, or children will not be eligible.
13. Psychiatric, other medical illness or other condition that in the opinion of the PI prevents compliance with study procedures or ability to provide valid informed consent
14. Use of anti-coagulant agents or history a significant bleeding diathesis. If a superficial lymph node or subcutaneous mass is to be injected, patients on agents such as non-steroidal anti-inflammatory drugs (NSAIDs), aspirin, or clopidogrel are eligible and these agents do not have to be withheld. For procedures with moderate or significant risk of bleeding, long-acting agents such as aspirin or clopidogrel should be discussed with the Sponsor and may need to be discontinued before Selicrelumab therapy. Patients under preventive dose of low molecular weight heparin (LMWH) are eligible if they can stop their treatment 24h prior the IT injection and restart 24h after the injection. No anticoagulant restriction for patients with injected lesions being superficial tumor lesions eligible for at least 5mn mechanical compression after tumor biopsy & injections (as in routine interventional radiology practice).
15. Subcapsular liver tumor lesions of tumor encased vessels or not eligible for intratumoral biopsies or injections.
16. Treatment with a live, attenuated vaccine within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during Atezolizumab treatment or within 5 months after the last dose of Atezolizumab
17. Prior allogeneic hematopoietic stem cell transplantation
18. Patients who have undergone a solid organ transplant
19. Documented infection with HIV
20. Positive serology to hepatitis B. Patients with previous and cured infections are not eligible. Patients who are seropositive due to a history of hepatitis B vaccine are eligible.
21. History or presence of an abnormal ECG that is clinically significant in the investigator's opinion, including complete left bundle branch block, second- or third degree heart block, or evidence of prior myocardial infarction
22. Person deprived of his/her liberty by a judicial or administrative decision
23. Person hospitalized without consent
24. Adult person under legal protection
25. Adult person unable to provide informed consent because of intellectual impairment, any serious medical condition, laboratory abnormality or psychiatric illness
26. Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-04-07 (Actual)

PRIMARY OUTCOMES:
optimal dose of intratumoral Selicrelumab in combination with flat doses of Atezolizumab IV | 21 days (1 cycle)

SECONDARY OUTCOMES:
complete metabolic response rate (CMR) | 2 months
complete metabolic response rate (CMR) | 4 months
complete metabolic response rate (CMR) | 8 months
complete metabolic response rate (CMR) | 13 months
overall metabolic response rate (OMR) | 2 months
overall metabolic response rate (OMR) | 4 months
overall metabolic response rate (OMR) | 8 months
overall metabolic response rate (OMR) | 13 months
Best overall metabolic response (BOMR) | 4 months
duration of response (DOR) | 2 years
progression free survival (PFS) | 2 years
overall survival (OS) | 2 years
Number of serious adverse event (SAE) | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Roch HOUOT, Pr, Study Chair — CHU Rennes
Locations (5):
- France (5):
  - APHP - Hôpital Henri Mondor, Créteil
  - CHU de Montpellier, Montpellier
  - Hospices Civils de Lyon - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Rennes - Hôpital Pontchaillou, Rennes
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No